CLINICAL TRIAL: NCT06754566
Title: A Caregiver-Assisted Rehabilitation With Strategy Training (CAR-ST) for Stroke Patients With Functional Limitations: A MultiCenter, 3-Arm Randomized Trial
Brief Title: A Caregiver-Assisted Rehabilitation With Strategy Training (CAR-ST) for Stroke Patients
Acronym: CAR-ST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Feng-Hang Chang, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202403026
Record Dates: First submitted 2024-12-30; First posted 2025-01-01 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Stroke; Caregiver-assisted rehabilitation; Strategy training; Activity limitations
MeSH Terms: conditions — Stroke | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: A researcher is responsible for the randomization process and the results are coded with predefined IDs that investigators and outcomes assessors are unaware of the meaning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caregiver-Assisted Rehabilitation with Strategy Training (CAR-ST) (Experimental): Trained therapists visit each participant once or twice weekly for 60 minutes. The program consists of 10 therapist-guided sessions over a maximum of 6 weeks and includes the following active ingredients: self-selected activity-based goals, dynamic performance analysis, global strategy ("Goal-PlanDo-Check"), massed practice, variable practice, increasing task difficulty, explicit and implicit feedback, guided discovery, action observation, and social interaction.
  Interventions: Behavioral: Caregiver-Assisted Rehabilitation with Strategy Training
- Strategy Training (Active Comparator): Participants assigned to the ST group receive a protocol similar to CAR-ST, with the distinction that their caregivers are not asked to co-participate in the intervention, and they are not instructed (by the research therapist) to provide assistance during at-home practice.
  Interventions: Behavioral: Strategy Training
- Education (Placebo Comparator): In this arm, participants receive a dose-matched intervention with 10 visits by well-trained research therapists through face-to-face talks (primary approach), video conference, or telephone calls. Sessions focus on instruction on general information regarding stroke and rehabilitation, and a summary of participants' condition and progression is provided for each visit.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Caregiver-Assisted Rehabilitation with Strategy Training — CAR-ST is a home-based rehabilitation that guides both stroke survivors and their caregivers to implement strategy training for addressing daily activity limitations after stroke. The caregiver, as an active partner, not only supervises the participant but also co-participates in the practice. Caregivers are instructed on when and how to provide assistance during task practice, using physical, verbal, or visual guidance. As the participant's performance improves, the caregiver is empowered to motivate them to exert greater efforts, encouraging higher repetitions, longer durations of the same task, and an increased level of difficulty.
  Other Names: CAR-ST
  Arms: Caregiver-Assisted Rehabilitation with Strategy Training (CAR-ST)
Behavioral: Strategy Training — Compared to CAR-ST, ST is a home-based rehabilitation that guides stroke survivors only to implement strategy training for addressing daily activity limitations after stroke.
  Other Names: ST
  Arms: Strategy Training
Behavioral: Education — Stroke-related information and knowledge that includes stroke subtypes and their etiology, risk factors of primary and secondary stroke, healthy lifestyles, common sequala, and adaptive skills for impaired functions are provided.
  Arms: Education

SUMMARY:
The goal of this randomized controlled trial is to examine if involving the caregivers in the strategy training (i.e. caregiver-assisted rehabilitation with strategy training, CAR-ST) works to improve activity functions in community-dwelling adults after stroke. The main questions it aims to answer are:

Does CAR-ST and strategy training alone lead to greater improvements in activity performance among stroke survivors relative to the control intervention with education? Does CAR-ST outperform strategy training alone in the efficacy of activity outcomes? Do the activity effects of CAR-ST transfer to the impairment and participation domains of outcomes?

Researchers will compare the efficacy of the CAR-ST intervention against strategy training alone or control intervention (education program) to see if caregivers contribute to post-stroke functional improvements.

Participants will:

* receive CAR-ST, strategy training only, or an education program 1 to 2 sessions per week until finishing 10 sessions.
* be assessed clinical outcomes at 4 times: pre-intervention, post-intervention, 3-month, and 6-month follow-up.

DETAILED DESCRIPTION:
Stroke is the leading cause of enduring disability worldwide, contributing to widespread impairments in survivors, thereby impeding various activities of daily life. Despite the effectiveness of intensive inpatient rehabilitation in mitigating deficits and activity limitations, maintaining an optimal treatment dose for patients transitioning to home remains a challenge. To address this gap, the integration of caregivers into home-based, evidence-supported rehabilitation emerges as a promising approach, yet its efficacy requires comprehensive examination. This clinical trial aims to assess the efficacy of a newly developed intervention, caregiver-assisted rehabilitation with strategy training (CAR-ST), in enhancing the activity performance of stroke survivors.

A single-blinded, three-arm randomized controlled trial will be executed, comparing the efficacy of the CAR-ST intervention against strategy training alone or attentional control through education. A procedure of randomization with minimization will be conducted by a researcher who is independent of the investigation and outcome assessments. Eligible stroke survivors and their caregivers will be recruited from collaborative hospitals in Northern Taiwan and randomly assigned with even possibility. Longitudinal evaluations will be conducted at baseline (T1), post-intervention (T2), 3-month (T3), and 6-month (T4) follow-ups, utilizing the Activity Measure for Post-Acute Care (AM-PAC) outpatient shortform as the primary outcome. Secondary outcomes will include the Participation Measure-3 Domains, 4 Dimensions (PM-3D4D), EuroQol-5D (EQ-5D), Stroke Self-Efficacy Questionnaires (SSEQ), Fugl-Meyer Assessment (FMA), Montreal Cognitive Assessment (MoCA), and Goal Attainment Scaling (GAS). Under the principles of modified intention-to-treat, quantitative data will be analyzed using multiple linear regression models and mixed-effects regression models. If data is lost at follow-up, inferential statistical analyses for group comparisons will be conducted both with or without multiple imputation. Furthermore, qualitative in-depth interviews with participants, caregivers, and therapists will be conducted post-intervention. These interviews will explore experiences, satisfaction, and perceived effectiveness of the intervention. Transcribed data will undergo coding by two independent coders and subsequent analysis through the thematic analysis method.

ELIGIBILITY:
Inclusion Criteria:

* Being willing to provide informed consent
* Diagnosis with ischemic and/or hemorrhagic stroke
* Modified Rankin Scale (mRS) ranges from 2 to 4
* Rehabilitation frequency less than 3 days per week
* Having a healthy caregiver

Exclusion Criteria:

* Undergoing palliative care
* Major diseases or severe conditions influencing study participation, such as global aphasia, dementia, multiple organ failure, immobilization due to fracture, etc
* Moderate post-stroke cognitive impairment, with Montreal Cognitive Assessment score <22
* Pre-stroke mRS > 1
* Participating in other interventional study concurrently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Activity Measure for Post-Acute Care (AM-PAC) Outpatient Short Forms | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  The AM-PAC measures the difficulty is performing three activity domains: Basic Mobility (18 activities), Daily Activity (15 activities), and Applied Cognition (19 activities) on a 4-point scale. In this trial, Applied Cognition domain is viewed as a secondary outcome. A trained research assistant performs AM-PAC face-to-face with participants.

SECONDARY OUTCOMES:
Participation Measure-3 Domains, 4 Dimensions (PM-3D4D) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  PM-3D4D consists of 24 items for evaluating three domains of participation, which are community, productivity, and social. Participants will be asked to rate all items on the four distinct dimensions: (1) diversity, (2) frequency, (3) desire for change, and (4) perceived difficulty. A trained research assistant performs PM-3D4D face-to-face with participants.
EuroQol-5D-3L (EQ-5D-3L) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  EuroQol-5D-3L (EQ-5D-3L) is a self-reported measurement that assesses participants' health-related quality of life across five domains: mobility, self-care, usual activity, pain/discomfort, anxiety/depression. In each domain, the assessment utilizes three levels to indicate the extent of problem: no problem, moderate problems, and extreme problems. A trained research assistant performs EQ-5D-3L face-to-face with participants.
Stroke Self-Efficacy Questionnaires (SSEQ) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  SSEQ measures individual confidence in functional performance after stroke [64]. It contains 13 items, and each item is rated on a 10-point scalar from 0 (not at all confident) to 10 (very confident). A trained research assistant performs SSEQ face-to-face with participants.
Fugl-Meyer Motor Assessment (FMA) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  FMA measures the motor impairments of hemiplegia and includes a proximal subscale of upper extremity (0-42 points) for the shoulder/elbow/forearm, distal subscale of upper extremity (0-24 points) for the wrist/hand, and a lower extremity subscale (0-34 points) A trained research assistant performs FMA face-to-face with participants.
Montreal Cognitive Assessment (MoCA) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  MoCA with 30 items evaluates the cognitive functions (range: 0-30). This assessment covers domains such as visuospatial/executive skills, naming, memory, attention, language, abstraction, delayed recall, and orientation. A trained research assistant performs MoCA face-to-face with participants.
Goal Attainment Scale (GAS) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  GAS is used to quantify the achievement of goals (range -3 to 2 for each goal). A trained research assistant performs GAS face-to-face with participants.

OTHER OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | At baseline, within 4 weeks after enrollment
  NIHSS is used to indicate participants' stroke severity before intervention (range 0-42).
modified Rankin Scale (mRS) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  mRS is used to indicate participants' global disability (0-6).
Berg Balance Scale (BBS) | At baseline, within 4 weeks after enrollment
  BBS is used to indicate participants' balance function before intervention (0-56).
Hospital Anxiety and Depression Scale (HADS) | At baseline, within 4 weeks after enrollment
  HADS is used to indicate participants' mood status before intervention (0-21).

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Heng Chang, ScD, Principal Investigator — Graduate Institute of Injury Prevention and Control, Taipei Medical University
Locations (5):
- Taiwan (5):
  - Taipei Tzu Chi Hospital, New Taipei City
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided